CLINICAL TRIAL: NCT00759161
Title: A Double-Blind, Randomized Bilateral Study of the Safety and Efficacy of AN2728 Ointment, 5%, Versus Ointment Vehicle in the Treatment of Patients With Plaque Type Psoriasis
Brief Title: Safety and Efficacy Study of A Novel Ointment to Treat Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN2728-PSR-201; C3291014 (Other: Pfizer)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Psoriasis
Keywords: Plaque Type Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): AN2728 Ointment, 5%
  Interventions: Drug: AN2728
- 2 (Placebo Comparator): AN2728 Ointment Vehicle
  Interventions: Drug: AN2728 Ointment Vehicle

INTERVENTIONS:
Drug: AN2728 — AN2728 Ointment, 5%, twice daily for 4 weeks
  Other Names: AN2728 Ointment, 5%
  Arms: 1
Drug: AN2728 Ointment Vehicle — AN2728 Ointment Vehicle, twice daily for 4 weeks.
  Arms: 2

SUMMARY:
The purpose of the study is to determine the safety and efficacy of AN2728 Ointment, 5%, compared to Ointment Vehicle in the treatment of plaque type psoriasis.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind bilateral design. Patients will apply the test articles, AN2728 Ointment, 5%, and Ointment Vehicle twice daily. The assigned study medication will be applied to two comparable treatment targeted plaques identified at baseline. One test article will be applied to one plaque and the other test article to an anatomically distinct plaque. All efficacy evaluations will be measured from only the two plaques identified at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at time of enrollment.
2. The clinical diagnosis of stable plaque psoriasis.
3. Two target plaques of similar severity

   1. ≥ 5 cm2 but ≤ 100 cm2 computed by multiplying the greatest diameter of the plaque by the diameter of the plaque perpendicular to the greatest diameter.
   2. Bilaterally located (right/left) plaques on the arms or plaques located on the upper and lower trunk. Plaques located on the trunk were to be separated by at least 10 cm and designated by the Investigator as either left/right or front/back.
   3. Target plaque severity score of 2-4 (mild to moderate).
4. Normal or not clinically significant screening laboratory results.
5. Subjects who were willing and able to apply study drug as directed, comply with study instructions, and commit to all follow-up visits.
6. Subjects who had the ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol related procedures.

Exclusion Criteria:

1. Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the patient to an unacceptable risk by study participation
2. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see below)
3. Known sensitivity to any of the components of the study medication
4. Spontaneously improving or rapidly deteriorating psoriatic plaques or pustular/exfoliative, guttate, erythrodermic or other non-plaque form of psoriasis
5. Concomitant use of topical or systemic therapies that might alter the course of psoriasis
6. Females of child bearing potential. Females must be post-menopausal (based on FSH levels) or surgically sterile (oophorectomy)
7. Washout periods of:

   1. Topical drugs that might alter the course of psoriasis: 2 weeks
   2. Oral retinoids: 8 weeks
   3. Non-retinoid systemic drugs that might alter the course of psoriasis: 4 weeks
   4. PUVA: 4 weeks
   5. UVB therapy: 4 weeks
   6. Use of emollients/moisturizers on area(s) to be treated: 2 days prior to baseline visit
8. AIDS or AIDS related illness
9. Concurrent participation in another drug research study or within 30 days of enrollment
10. Use of lithium or hydroxychloroquine containing products (i.e. Plaquenil)
11. Use of a beta-blocking medication (i.e. propranolol) if the dose has not been stabilized for at least 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- IMIC, Mexico City, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 5% Ointment + Ointment Vehicle: AN2728 ointment, 5 percent (%) and ointment vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques within each participant respectively, twice daily for 4 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (9.03)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Decrease in Overall Target Plaque Severity Score (OTPSS) at Day 28
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored on a severity rating scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicated more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS at Day 28 were reported and comparison of ointment and vehicle treated plaque was given as 'Ointment treated plaque versus (vs.) vehicle treated plaque' and 'Vehicle treated plaque vs. ointment treated plaque'.
Time Frame: Day 28
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 35
percentage of participants
  Ointment treated plaque vs. vehicle treated plaque | 68.6
  Vehicle treated plaque vs. ointment treated plaque | 5.7
Statistical Analysis 1: Comparison: AN2728 5% Ointment + Ointment Vehicle; Test type: Superiority or Other; p < 0.001, 2-sided sign test

2. Secondary Outcome: Change From Baseline in Overall Target Plaque Severity Score (OTPSS) at Day 7,14, 21, 28 and 35
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored on a severity scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicated more severity of a plaque.
Time Frame: Baseline (Day 1), Day 7,14, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AN2728 5% Ointment: AN2728 ointment, 5 percent (%) was applied to 1 of the 2 comparable and anatomically distinct treatment-targeted plaques within each participant, twice daily for 4 weeks. Plaques were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment Vehicle: AN2728 ointment vehicle was applied to 1 of the 2 comparable and anatomically distinct treatment-targeted plaques within each participant, twice daily for 4 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 5% Ointment | AN2728 Ointment Vehicle
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline | 2.8 (0.53) | 2.8 (0.53)
  Change at Day 7 | 0.17 (0.453) | 0.11 (0.404)
  Change at Day 14 | 0.71 (0.572) | 0.31 (0.583)
  Change at Day 21 | 1.06 (0.539) | 0.49 (0.658)
  Change at Day 28 | 1.40 (0.497) | 0.66 (0.684)
  Change at Day 35 | 1.26 (0.505) | 0.57 (0.655)

3. Secondary Outcome: Change From Baseline in Erythema at Day 7,14, 21, 28 and 35
Description: Erythema is used to assess plaque severity. Investigator rated the clinical appearance of erythema on a severity scale, ranging from 0 (no color on plaque, no erythema) to 8 (extreme red color on plaque, severe erythema), where higher score indicated more severe condition.
Time Frame: Baseline (Day 1), Day 7,14, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ointment Vehicle: AN2728 ointment vehicle was applied to 1 of the 2 comparable and anatomically distinct treatment-targeted plaques within each participant, twice daily for 4 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 5% Ointment | Ointment Vehicle
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline | 2.8 (0.62) | 2.8 (0.57)
  Change at Day 7 | 0.31 (0.631) | 0.14 (0.430)
  Change at Day 14 | 0.63 (0.731) | 0.29 (0.622)
  Change at Day 21 | 1.09 (0.658) | 0.40 (0.695)
  Change at Day 28 | 1.40 (0.651) | 0.60 (0.736)
  Change at Day 35 | 1.37 (0.770) | 0.57 (0.778)

4. Secondary Outcome: Change From Baseline in Scaling at Day 7,14, 21, 28 and 35
Description: Scaling is a scale to assess plaque severity. Investigator rated the clinical appearance of scaling on a severity scale, ranging from 0 (no scaling on plaque) to 8 (very thick scales on plaque), where higher score indicated more severe condition.
Time Frame: Baseline (Day 1), Day 7,14, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 5% Ointment | Ointment Vehicle
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline | 3.2 (0.73) | 3.1 (0.63)
  Change at Day 7 | 0.69 (0.676) | 0.43 (0.502)
  Change at Day 14 | 1.29 (0.667) | 0.89 (0.631)
  Change at Day 21 | 1.60 (0.812) | 0.94 (0.725)
  Change at Day 28 | 1.83 (0.747) | 1.09 (0.818)
  Change at Day 35 | 1.66 (0.838) | 0.91 (0.742)

5. Secondary Outcome: Change From Baseline in Plaque Elevation at Day 7,14, 21, 28 and 35
Description: Plaque elevation is a scale to assess plaque severity. Investigator rated presence of plaque elevation on a severity scale ranging, from 0 (no plaque elevation) to 8 (very marked plaque elevation), where higher score indicated more severe condition.
Time Frame: Baseline (Day 1), Day 7,14, 21, 28, 35
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 5% Ointment | Ointment Vehicle
Number analyzed (Participants) | 35 | 35
units on a scale
  Baseline | 2.7 (0.61) | 2.7 (0.58)
  Change at Day 7 | 0.17 (0.453) | 0.03 (0.296)
  Change at Day 14 | 0.49 (0.562) | 0.26 (0.611)
  Change at Day 21 | 0.83 (0.707) | 0.26 (0.611)
  Change at Day 28 | 1.23 (0.731) | 0.40 (0.604)
  Change at Day 35 | 1.20 (0.632) | 0.43 (0.655)

6. Secondary Outcome: Percentage of Participants With Greater Decrease in Overall Target Plaque Severity Score (OTPSS) at Day 7,14, 21 and 35
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored on a severity rating scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicated more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS at Day 7, 14, 21 and 35 were reported and comparison of ointment and vehicle treated plaque was given as 'Ointment treated plaque vs. vehicle treated plaque' and 'Vehicle treated plaque vs. ointment treated plaque'.
Time Frame: Day 7,14, 21, 35
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 35
percentage of participants
  Day 7: Ointment treated vs.vehicle treated plaque | 11.4
  Day 7: Vehicle treated vs.ointment treated plaque | 5.7
  Day 14: Ointment treated vs.vehicle treated plaque | 48.6
  Day 14: Vehicle treated vs.ointment treated plaque | 8.6
  Day 21:Ointment treated vs.vehicle treated plaque | 54.3
  Day 21: Vehicle treated vs.ointment treated plaque | 2.9
  Day 35:Ointment treated vs.vehicle treated plaque | 62.9
  Day 35: Vehicle treated vs.ointment treated plaque | 2.9

ADVERSE EVENTS:
Groups:
- AN2728 5% Ointment + Ointment Vehicle: AN2728 ointment, 5 percent (%) and ointment vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques within each participant, twice daily for 4 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 5% Ointment + Ointment Vehicle (N=35)
Diarrhoea (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.